CLINICAL TRIAL: NCT05071729
Title: Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Elinzanetant in Participants With Impaired Renal Function in Comparison to Matched Controls With Normal Renal Function
Brief Title: A Study to Learn How Elinzanetant Moves Into, Through, and Out of the Body, How Safe it is, and How it Affects the Body in Participants With Kidneys That do Not Work as Well as They Should Compared to Participants Whose Kidneys Work Normally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21669
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
Keywords: Hot flushes; Elinzanetant; Investigation of pharmacokinetics and safety in renal impaired participants
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate renal impairment (Experimental): Participants with estimated glomerular filtration rate (eGFR) of 30 to 59 mL/min/1.73 m^2
  Interventions: Drug: Elinzanetant (BAY3427080)
- Severe renal impairment (Experimental): Participants with eGFR < 30 mL/min/ 1.73 m^2
  Interventions: Drug: Elinzanetant (BAY3427080)
- Normal renal function (Experimental): Participants with ≥ 90 mL/min/1.73 m^2
  Interventions: Drug: Elinzanetant (BAY3427080)

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Single oral dose of elinzanetant on Day 1.

SUMMARY:
Researchers are looking for a better way to treat people who have vasomotor symptoms (VMS).

The symptoms of VMS are hot flashes. These symptoms can be caused by changes in sex hormone levels. An example of a change in sex hormone levels is when a woman reaches the time in their life where they no longer have their period. Hormones are substances in the blood that help body organs to work in specific ways. Women who no longer have their period may have a protein called neurokinin sending more signals than usual to other parts of the body. Researchers think that this may play a role in causing VMS.

In this study, the researchers want to learn more about a new substance called elinzanetant. Researchers think elinzanetant may help people with VMS. It works by blocking neurokinin from sending signals to other parts of the body. There are treatments available for VMS, but these do not work for all people and may cause medical problems for some people.

The main purpose of this study is to help the researchers learn more about how elinzanetant moves into, through and out of the body in participants with kidneys that do not work as well as they should compared to healthy participants whose kidneys work normally. To do this, the doctors will take blood samples from the participants at different times during the study and measure the levels of elinzanetant in the blood. This will help the researchers learn more about whether elinzanetant could be given to treat VMS in people who also have kidneys that do not work as well as they should.

This study will include adult participants who have kidneys that do not work as well as they should and participants whose kidneys work normally. The participants who have kidneys that do not work as well as they should will be split into 2 groups based on how severe their kidney problems are. All of the participants will take elinzanetant once as a tablet by mouth.

The participants will be in the study for about 1 month and will stay at their study site for 7 days in a row. During this visit, the participants will:

* have their overall health checked
* have scans of their heart taken using an electrocardiogram
* have blood and urine samples taken
* answer questions about how they are feeling, what medications they are taking, and what adverse events they are having

The doctors will keep track of any adverse events. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent.
* Moderate or severe renal impairment as assessed by estimated glomerular filtration rate (eGFR) based on serum creatinine collected 2 to 10 days prior to dosing and calculated according to a modified Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI). Moderately impaired renal function: eGFR: 30 up to 59 mL/min/1.73 m^2 (inclusive); Severely impaired renal function: eGFR < 30 mL/min/ 1.73 m^2 (including at least 50% patients requiring hemodialysis).
* Stable renal disease, i.e. a serum creatinine value determined 3 or more months before screening (e.g. during routine diagnostics) should not differ by more than 25% from the serum creatinine value determined at screening.
* Normal renal function, as assessed by eGFR based on serum creatinine at screening according to the modified CKD-EPI formula: eGFR ≥90 mL/min/1.73 m^2.
* Body mass index (BMI) within the range 18 - 32 kg/m^2 (inclusive).
* Male or female.
* Study participants of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period from signing of the informed consent form (ICF) until the follow-up visit on Day 6. Use of adequate contraception should be consistent with local regulations.

Exclusion Criteria:

* Any relevant disease (other than those related to renal impairment for the renal impaired participants) within 4 weeks prior to study drug administration including infections and acute gastro-intestinal diseases (with vomiting, diarrhea, constipation, etc.) requiring medical treatment.
* Acute renal failure or acute nephritis within the past 2 years.
* Malignancy diagnosed or treated within the past 5 years (hepatocellular carcinoma within the past 2 years). This does not include adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin.
* Conditions associated with a risk of hypersensitivity reactions with study intervention (active substances, or excipients of the preparations) as judged by the investigator.
* Dialysis for acute renal failure within the previous 6 months prior to administration of study intervention.
* Use of drugs which may affect absorption (e.g. loperamide, metoclopramide),and systemic administration of any broad-spectrum antibiotic within 1 week before study drug administration, unless the drug is part of the mandatory dosing regimen for treatment of renal impairment or related conditions.
* Use of drugs which may affect absorption by increasing the gastro-intestinal pH e.g. proton pump inhibitors from 2 weeks before study drug administration until last day of blood sampling for PK after study drug administration.
* Use of anti-coagulant drugs other than 100 mg acetylsalicylic acid per day.
* Major change of any medication regimen less than 2 weeks prior to first study drug administration, including dose adjustments.
* Indication for immunosuppressants, receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy within 6 months prior to administration of study intervention
* Women of childbearing potential with a positive pregnancy test at screening or on Day -1.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve in plasma from zero to infinity (AUCu) (unbound) | Predose up to 120 hours
  Measured matrix after a single dose administration.
Maximum observed (unbound) drug concentration (Cmax,u) | Predose up to 120 hours
  Maximum observed (unbound) drug concentration (Cmax,u) in measured matrix after a single dose administration.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events, categorized by severity | After administration of study intervention up to the follow-up visit on Day 6.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21669